CLINICAL TRIAL: NCT00828087
Title: A Clinical Evaluation of Everolimus Eluting Coronary Stents in the Treatment of Patients With ST-segment Elevation Myocardial Infarction.EXAMINATION Study
Brief Title: A Clinical Evaluation of Everolimus Eluting Coronary Stents in the Treatment of Patients With ST-segment Elevation Myocardial Infarction: EXAMINATION Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spanish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Dr. Sabate, Doctor, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EXAM-08
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Myocardial Infarction
Keywords: acute myocardial infarction; primary percutaneous coronary intervention; drug-eluting stent
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everolimus Arm (Experimental): Everolimus Eluting Coronary Stent System
  Interventions: Drug: Everolimus Eluting Coronary Stent System
- non drug eluting stent Arm (Active Comparator): cobalt chromium balloon expandable stent
  Interventions: Device: cobalt chromium balloon expandable stent ( non drug eluting stent Arm)

INTERVENTIONS:
Drug: Everolimus Eluting Coronary Stent System — Everolimus Eluting Coronary Stent System (Everolimus Arm) implantation
  Other Names: N/H
  Arms: Everolimus Arm
Device: cobalt chromium balloon expandable stent ( non drug eluting stent Arm) — cobalt chromium balloon expandable stent ( non drug eluting stent Arm)implantation
  Other Names: N/H.
  Arms: non drug eluting stent Arm

SUMMARY:
This study is a prospective, randomized controlled, single blind, two-arm, multi center clinical evaluation. A total of 1500 patients will be enrolled in the study.

Patient randomization will be to one of the two treatment arms: Everolimus arm or Non drug eluting stent arm. The objective of this study is to assess the safety and performance of the Everolimus Eluting Coronary Stent System versus a modified cobalt chromium balloon expandable stent in the setting of primary percutaneous coronary intervention for treatment of patients presenting with ST-segment elevation myocardial infarction.

DETAILED DESCRIPTION:
Primary PCI, with or without stenting, has been shown to result in superior long-term outcome when compared to thrombolytic therapy in patients with acute myocardial infarction (MI).

Recently, several studies showed that both sirolimus- and paclitaxel-eluting stents are more effective in reducing restenosis and the frequency of repeat interventions than bare metal stents, which rapidly resulted in an unrestricted use of drug-eluting stents, also in patients with ST segment elevation MI (STEMI). , , , Shortly after the introduction of the sirolimus-eluting stent in April 2002 the first studies appeared, hypothesizing that the therapeutic range of sirolimus-eluting stents could be extended to patients presenting with MI. When compared to bare metal stents, sirolimus-eluting stents were associated with less restenosis and target vessel revascularization (TVR) up until one year of follow-up. , At present, it is unclear whether this also holds for paclitaxel-eluting stents.4,

Everolimus is a sirolimus analogue, an effective anti-proliferative agent that inhibits growth factor-stimulated cell proliferation by causing cell cycle arrest in the late G1 stage in the cell cycle.

The objective of this study is to assess the safety and performance of the Everolimus Eluting Coronary Stent System versus a modified cobalt chromium balloon expandable stent in the setting of primary percutaneous coronary intervention for treatment of patients presenting with ST-segment elevation myocardial infarction.

This study is a prospective, randomized controlled, single blind, two-arm, multi center clinical evaluation. A total of 1500 patients will be enrolled in the study.

The primary endpoint is the combined endpoint of Composite endpoint of all-cause death, any myocardial infarction and any revascularization at 1 year (patient oriented endpoint suggested by the ARC definitions).

The following secondary endpoints will be examined:

* All cause and cardiac mortality at 1 year and yearly up to 5 years.
* Recurrent myocardial infarction at 1 year and yearly up to 5 years.
* Target lesion revascularization at 1 year and yearly up to 5 years.
* Target vessel revascularization at 1 year and yearly up to 5 years.
* Stent thrombosis (according to the new definitions proposed by the Academic Research Consortium) at 1 year and yearly up to 5 years.
* Clinical device success
* Clinical procedure success.
* Major and minor bleeding at 1 year and yearly up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with a ST-elevation myocardial infarction who must meet at least one of the following criteria

  * Patients presenting with a ST-elevation myocardial infarction <12 hours after onset of symptoms who are treated with primary angioplasty + stent implantation
  * Cardiogenic shock.
  * Rescue PCI after failed thrombolysis.
  * PCI indicated early (<24h) after effective thrombolysis following current ESC guidelines.
  * Patients presenting late ("latecomers") with ST-elevation myocardial infarction (>12h-48h) after the onset of symptoms.
* Written informed consent.
* The patient or his/her family (in the event the patient can not be clinically available) accept clinical controls.

Angiographic:

* Vessel size has to range between 2.25-4.0 mm by visual estimation to allow the implantation of currently available stents.

Exclusion Criteria:

* Age < 18 years.
* Pregnancy or breastfeeding.
* Known intolerance to aspirin, clopidogrel, heparin, stainless steel, Everolimus, contrast material.
* Patients with absolute indication of being chronic treated with acenocoumarol
* Myocardial infarction due to a previously implanted stent thrombosis
* Patients with myocardial infarction that will require elective surgical coronary revascularisation within a 1 year period (example: inferior MI with severe disease in left main with surgical indication).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1504 (Actual)
Dates: Start 2008-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of all-cause death, any myocardial infarction and any revascularization at 1 year. | 1 year

SECONDARY OUTCOMES:
All cause and cardiac mortality | at 1 year and yearly up to 5 years
Recurrent myocardial infarction | at 1 year and yearly up to 5 years
Target lesion revascularization | at 1 year and yearly up to 5 years
Target vessel revascularization | at 1 year and yearly up to 5 years
Stent thrombosis | at 1 year and yearly up to 5 years
Clinical device success | Procedure moment
  Successful delivery and deployment of the first inserted stent and a final diameter stenosis after stenting ≤ 50% by QCA or visual assessment.
Clinical procedure success | procedure moment
  Successful delivery and deployment of study stent in the target lesion and successful removal of the stent delivery system with a final diameter stenosis after stenting ≤ 50% by QCA or visual assessment without the occurrence of serious cardiac events important for ischemia during hospitalization, with a maximum of seven days after the initial procedure.
Major and minor bleeding | at 1 year and yearly up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Prof. P.W. Serruys, MD,PhD, Principal Investigator — Erasmus MC, Rotterdam; Manuel Sabate, MD,PhD, Principal Investigator — Hospital Clínic i Provincial de Barcelona
Locations (11):
- Italy (2):
  - Azienda Ospedaliera Bolognini, Seriate, Bergamo
  - Azienda Ospedaliero Universitaria S. Anna di Ferrara, Ferrara, Italy
- Erasmus MC, Rotterdam, Rotterdam, Rotterdam, Netherlands
- Spain (8):
  - Complejo Hospitalario U. A Coruña, A Coruña, A Croruña
  - Hospital General de Alicante, Alicante, Alicante
  - Hospital Son Dureta, Palma de Mallorca, Balearic Islands
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona, Barcelona
  - Hospital de Bellvitge, Barcelona, Barcelona
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital do Meixoeiro, Vigo, Vigo

REFERENCES:
- [Derived] Costa F, Brugaletta S, Pernigotti A, Flores-Ulmanzor E, Ortega-Paz L, Cequier A, Iniguez A, Serra A, Jimenez-Quevedo P, Mainar V, Campo G, Tespili M, den Heijer P, Bethencourt A, Vazquez N, van Es GA, Backx B, Valgimigli M, Serruys P, Sabate M. Does Large Vessel Size Justify Use of Bare-Metal Stents in Primary Percutaneous Coronary Intervention? Circ Cardiovasc Interv. 2019 Sep;12(9):e007705. doi: 10.1161/CIRCINTERVENTIONS.118.007705. Epub 2019 Aug 27. PMID 31451013
- [Derived] Schur N, Brugaletta S, Cequier A, Iniguez A, Serra A, Jimenez-Quevedo P, Mainar V, Campo G, Tespili M, den Heijer P, Bethencourt A, Vazquez N, Valgimigli M, Serruys PW, Ademi Z, Schwenkglenks M, Sabate M. Cost-effectiveness of everolimus-eluting versus bare-metal stents in ST-segment elevation myocardial infarction: An analysis from the EXAMINATION randomized controlled trial. PLoS One. 2018 Aug 16;13(8):e0201985. doi: 10.1371/journal.pone.0201985. eCollection 2018. PMID 30114230
- [Derived] Gomez-Lara J, Brugaletta S, Jacobi F, Ortega-Paz L, Nato M, Roura G, Romaguera R, Ferreiro JL, Teruel L, Gracida M, Martin-Yuste V, Freixa X, Masotti M, Gomez-Hospital JA, Sabate M, Cequier A. Five-Year Optical Coherence Tomography in Patients With ST-Segment-Elevation Myocardial Infarction Treated With Bare-Metal Versus Everolimus-Eluting Stents. Circ Cardiovasc Interv. 2016 Oct;9(10):e003670. doi: 10.1161/CIRCINTERVENTIONS.116.003670. PMID 27702766
- [Derived] Sabate M, Brugaletta S, Cequier A, Iniguez A, Serra A, Jimenez-Quevedo P, Mainar V, Campo G, Tespili M, den Heijer P, Bethencourt A, Vazquez N, van Es GA, Backx B, Valgimigli M, Serruys PW. Clinical outcomes in patients with ST-segment elevation myocardial infarction treated with everolimus-eluting stents versus bare-metal stents (EXAMINATION): 5-year results of a randomised trial. Lancet. 2016 Jan 23;387(10016):357-366. doi: 10.1016/S0140-6736(15)00548-6. Epub 2015 Oct 29. PMID 26520230
- [Derived] Taniwaki M, Stefanini GG, Raber L, Brugaletta S, Cequier A, Heg D, Iniguez A, Kelbaek H, Serra A, Ostoijic M, Hernandez-Antolin R, Baumbach A, Blochlinger S, Juni P, Mainar V, Sabate M, Windecker S. Predictors of adverse events among patients undergoing primary percutaneous coronary intervention: insights from a pooled analysis of the COMFORTABLE AMI and EXAMINATION trials. EuroIntervention. 2015 Aug;11(4):391-8. doi: 10.4244/EIJY14M07_12. PMID 25042419
- [Derived] Fernandez-Rodriguez D, Regueiro A, Brugaletta S, Martin-Yuste V, Masotti M, Cequier A, Iniguez A, Serra A, Hernandez-Antolin R, Mainar V, Valgimigli M, Tespili M, den Heijer P, Bethencourt A, Vazquez N, Serruys PW, Sabate M; EXAMINATION investigators. Optimization in stent implantation by manual thrombus aspiration in ST-segment-elevation myocardial infarction: findings from the EXAMINATION trial. Circ Cardiovasc Interv. 2014 Jun;7(3):294-300. doi: 10.1161/CIRCINTERVENTIONS.113.000964. Epub 2014 May 27. PMID 24867891
- [Derived] Sabate M, Brugaletta S, Cequier A, Iniguez A, Serra A, Hernadez-Antolin R, Mainar V, Valgimigli M, Tespili M, den Heijer P, Bethencourt A, Vazquez N, Backx B, Serruys PW. The EXAMINATION trial (Everolimus-Eluting Stents Versus Bare-Metal Stents in ST-Segment Elevation Myocardial Infarction): 2-year results from a multicenter randomized controlled trial. JACC Cardiovasc Interv. 2014 Jan;7(1):64-71. doi: 10.1016/j.jcin.2013.09.006. Epub 2013 Dec 11. PMID 24332423
- [Derived] Sabate M, Cequier A, Iniguez A, Serra A, Hernandez-Antolin R, Mainar V, Valgimigli M, Tespili M, den Heijer P, Bethencourt A, Vazquez N, Gomez-Hospital JA, Baz JA, Martin-Yuste V, van Geuns RJ, Alfonso F, Bordes P, Tebaldi M, Masotti M, Silvestro A, Backx B, Brugaletta S, van Es GA, Serruys PW. Everolimus-eluting stent versus bare-metal stent in ST-segment elevation myocardial infarction (EXAMINATION): 1 year results of a randomised controlled trial. Lancet. 2012 Oct 27;380(9852):1482-90. doi: 10.1016/S0140-6736(12)61223-9. Epub 2012 Sep 3. PMID 22951305
- [Derived] Sabate M, Cequier A, Iniguez A, Serra A, Hernandez-Antolin R, Mainar V, Valgimigli M, Tespili M, den Heijer P, Bethencourt A, Vazquez N, Brugaletta S, Backx B, Serruys P. Rationale and design of the EXAMINATION trial: a randomised comparison between everolimus-eluting stents and cobalt-chromium bare-metal stents in ST-elevation myocardial infarction. EuroIntervention. 2011 Dec;7(8):977-84. doi: 10.4244/EIJV7I8A154. PMID 22115622